CLINICAL TRIAL: NCT06930365
Title: Clinical-Instrumental Study To Evaluate And Compare The Efficacy And Tolerability Of Two Emollients Products (Investigational Product Versus Placebo) In Atopic Dermatitis
Brief Title: Clinical-Instrumental Study To Evaluate And Compare The Efficacy And Tolerability Of Two Emollients Products In Atopic Dermatitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NAOS Les Laboratoires (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC2024/PSaib+/GE
Record Dates: First submitted 2025-02-24; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Atopic Dermatitis; Eczema
Keywords: Eczema; Atopic Dermatisis; Body Cream
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — Diphenhydramine

STUDY DESIGN:
Intervention Model Description: Interventional , monocentric, double-blinded, randomized and comparative study. The study design is randomized: Enrolled participants will apply the new emollient versus placebo according to a previous defined randomization scheme.
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amr 1: New Emollient (Experimental): Study product, Emollient. Face and body
  Interventions: Other: Anti-itching and repairing treatment. Emollient.
- Arm 2: Placebo (Placebo Comparator): Product 2: Placebo, Emollient. face and body
  Interventions: Other: Emollient cream

INTERVENTIONS:
Other: Anti-itching and repairing treatment. Emollient. — Anti-itching and repairing treatment. Emollient.
  Arms: Amr 1: New Emollient
Other: Emollient cream — Emollient cream
  Arms: Arm 2: Placebo

SUMMARY:
Atopic dermatitis (AD) is a chronic inflammatory skin disease associated with erythema, scaly and oozing plaques, and severe pruritus which has an important impact on quality of life and quality of sleep. It is divided into 2 chronic phases : flare-up and remission period.

Signs and symptoms of AD are associated with a compromised immune system, a defective skin barrier, a cutaneous dysbiosis and overall inflammatory status.

The aim of the study is to evaluate and compare the efficacy and tolerability of two face and body cream products, new emollient versus placebo, in used over the course of 5 weeks as a replacement of usual or any emollient by female and male subjects with atopic dermatitis.

This is an interventional, single-center, double-blind, randomized and comparative study.

ELIGIBILITY:
Inclusion Criteria:

* Female and/or male participants,
* Participant aged between 18 years old and more included,
* All ethnicities
* Phototype II to IV
* Participant with all skin types, sensitive or not sensitive,
* 44 subjects having a rash of eczema (SCORAD between 25 and 50) with at least 1 lesional area requiring topical corticosteroid treatment,
* 22 healthy subjects (without any dermatological pathology nor disorder),
* 44 participants having whitened eczema lesions at Dx (between 5 to 10 days) after the topical corticosteroid treatment,
* Participants having signed their written Informed Consent form (ICF) for their participation in the study and a photograph authorization,
* Participant able to comply with the protocol and follow protocol's constraints and specific requirements.

Exclusion Criteria:

* Participant does not meet the inclusion criteria,
* Known pregnancy, participant breastfeeding, or not willing to take necessary precautions to avoid a pregnancy during the study,
* Participant with dermatological problems in the test areas other than atopic dermatitis,
* Pharmacological treatments (topic or systemic) other than topical corticosteroids, known to interfere with skin metabolism / physiology. In particular, no antibiotics taken within 4 weeks preceding the inclusion, nor anti- inflammatories taken within 2 weeks before the inclusion
* Participant being deprived of liberty by judicial or administrative decision, or under guardianship,
* Participant being linguistically or psychologically incapable of signing informed consent and unable to comply with the protocol requirements,
* Participant who has a relevant change in his state of health since registered in the LTD "Health" Database (change incompatible with inclusion in the study),
* Participant currently enrolled in another similar clinical study or in an exclusion period of a study,
* Participant having a skin recently exposed to sunlight (natural or artificial) and / or having applied a self-tanner on the application areas and /or tanning activator (dietary supplement) within 2 weeks preceding the inclusion.
* Participant having bathed in a swimming pool within 1 week preceding the inclusion or planning to bath in a swimming pool during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-05-16 (Estimated); Study Completion 2025-07-18 (Estimated)

PRIMARY OUTCOMES:
SCORAD (SCOring Atopic Dermatisis) | Day 0, Day 5 to Day 10, Day 5 to Day 10+28 (+/- 48 hours)
  SCORAD (SCOring Atopic Dermatisis). The SCORAD (Scoring Atopic Dermatitis) scale ranges from a minimum score of 0 to a maximum score of 103, where higher scores indicate a worse outcome, reflecting more severe atopic dermatitis.
EASI (Eczema Area and Severity Index) | Day 0, Day 5 to Day 10, Day 5 to Day 10+28 (+/- 48 hours)
  EASI (Eczema Area and Severity Index). The EASI (Eczema Area and Severity Index) ranges from 0 to 72, where higher scores indicate more severe atopic dermatitis, with 0 meaning no eczema and 72 representing the most severe form.
Transepidermal water loss by Vapometer® | Day 0, Day 5 to Day 10, Day 5 to Day 10+28 (+/- 48 hours)
  Transepidermal water loss by Vapometer® (on a defined AD lesion and on non-lesional area to the forearm))
Samplings of the cutaneous microbiota | Day 0, Day 5 to Day 10, Day 5 to Day 10+28 (+/- 48 hours)
  Samplings of the cutaneous microbiota on one or two defined AD lesion. If the subject presents 2 AD lesions, 2 microbiota samples will be done.
Filling of a DLQI questionnaires by participants | Day 0, Day 5 to Day 10, Day 5 to Day 10 + 28 (+/- 48hours)
  The DLQI (Dermatology Life Quality Index) ranges from 0 to 30, with higher scores indicating a greater impact of skin disease on quality of life. A score of 0-1 suggests no effect, while 30 indicates maximum impact.
Sleep quality by questionnaire (Pittsburgh Sleep Quality Index) filled in by participants | Day 0, Day 5 to Day 10, Day 5 to Day 10 + 28 (+/- 48hours)
  The Pittsburgh Sleep Quality Index (PSQI) ranges from 0 to 21, with higher scores indicating poorer sleep quality. A score above 5 suggests poor sleep, while a score of 0 indicates good sleep quality.
Safety Endpoints | Day 0, Day 5 to Day 10, Day 5 to Day 10 + 28 (+/- 48hours)
  Incidence, severity and causality of adverse events and serious adverse events
  Dermatological tolerance evaluation by clinical examination of the physical and functional signs done by a dermatologist
Safety Endpoints | Day 0, Day 5 to Day 10, Day 5 to Day 10 + 28 (+/- 48hours)
  Incidence, severity and causality of adverse events and serious adverse events
  Tolerance feedback by participants by Daily log (filled in by participants during the treatment period).
Safety Endpoints | Day 0, Day 5 to Day 10, Day 5 to Day 10 + 28 (+/- 48hours)
  Incidence, severity and causality of adverse events and serious adverse events
  Overall skin tolerance (skin reactions evaluated by the dermatologist and the ones reported by the participants) after 28 days of the tested product use determined by Dermatologist

CONTACTS AND LOCATIONS:
Locations (1):
- Ltd Health, Batumi, Adjara, Georgia